CLINICAL TRIAL: NCT04855838
Title: Impaired Swallowing Function After Anterior Cervical Spine Surgery- Incidence, Long-term Effect on Nutrition and Effect of Oral Neuromuscular Training
Brief Title: Dysphagia After Anterior Cervical Spine Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: University Hospital, Umeå (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019-06543
Record Dates: First submitted 2021-04-20; First posted 2021-04-22 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Dysphagia; Cervical Spinal Cord Injury
Keywords: Swallowing disorder; Anterior cervical spine surgery; Intervention; Incidens; Nutritional status
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): Intensive training with oral neuromuscular device (intervention group) and traditional compensatory swallowing training under 8 weeks with start 4 (±1) weeks post-operation.
  Interventions: Device: Oral neuromuscular training
- Control group (No Intervention): Traditional compensatory swallowing training under 8 weeks with start 4 (±1) weeks post-operation.

INTERVENTIONS:
Device: Oral neuromuscular training — The oral device is used for 30 seconds, three times a day, before meals and implies new possibilities for training of the orofacial and pharyngeal muscles.
  Arms: Intervention group

SUMMARY:
The purpose of this research project is to investigate the incidence of impaired swallowing (dysphagia) after anterior cervical spine surgery (ACSS) and to study the long-term effect of dysphagia on nutritional status 12 ± 3 months later. Furthermore, to investigate the effect of a new rehabilitation method for dysphagia among individuals with swallowing dysfunction after ACSS.

DETAILED DESCRIPTION:
Study design: This study contains of two parts. The first part of this study is a prospective observational cohort study with consecutive observations on the characterization of incidence of and factors related to dysphagia after ACSS (within 14 days of surgery and 2-3 weeks later), and investigation the long-term effect of dysphagia on nutritional status 12 ± 3 months later.

The second part of this study is a prospective randomized open-label trial with blinded evaluators (PROBE-design) that compare conventional care to neuromuscular training in the treatment of dysphagia.

Subjects and procedure: Part 1: All patients enrolled at the University Hospital of Umeå who have undergone ACSS between C2 and Th1 level due to trauma are eligible participants in the first part of the study (the observational cohort study). All participants will have their swallowing function assessed with a flexible video endoscopic evaluation of swallowing (i.e. FESS) within 14 days after surgery and have their nutritional status examined with the clinical test Nutrition Risk Screening-2002 (NRS-2002) and blood sample for biomarkers of malnutrition (i.e., levels of Albumin, levels of Leptin, Ghrelin and Adiponektin and also metabolites as ketone bodies (3 hydoxibutyrat and acetoacetate). The swallowing assessment and nutritional screening with NRS-2002 will be performed by a speech- language pathologist or physician in otolaryngology. Blood sample will be collected by a nurse at the unit where the participant is staying, who have extended knowledge in the procedure. If a swallowing dysfunction is present the patient will be followed-up within 2-3 weeks later (i.e., 4±1- week post-operation) to assess the spontaneous recovery. During the period from the first assessment to the follow-up all patients will be given conventional care (e.g., postural adjustments, swallowing maneuvers, modified consistency of solid and/or liquid food). If the patient has a remaining swallowing dysfunction at the reassessment 4±1-week post-operation the patient will be asked to participate in part 2 of the study (the interventional study). All patients participating in part 1, will have another examination of nutritional status at 12 ± 3 months after ACSS. In order to study the long-term effect of dysphagia on nutrition.

Part 2: Participants with presenting swallowing dysfunction at the reassessment 4±1 week post- operation will after given their oral or written consent be randomly assigned to 8 weeks of either conventional care (control group) or oral neuromuscular training with an oral device (intervention group). Randomization will be performed web-based using the program MINIM with minimization/ stratification for aspiration (yes/no) on FEES leading to an equal balance of prognostic important variable at baseline. In each group, swallowing function, swallowing-related quality of life measured by the Swallowing Quality of life Questionnaire (SWAL-QOL) and an examination of nutritional status with the clinical screening NRS-2002 and blood samples will be assessed at baseline (i.e. 4±1 week post-surgery assessment), eight weeks after baseline (end-of treatment), and 12 ± 3 months post-treatment. A swallowing assessment will also be performed four weeks into the treatment period. If oral neuromuscular training with an oral device is found to be effective in the intervention group, it will be also offered to the control group after the study is finished. All assessments will be carried out at the University Hospital of Umeå. All the assessments of the participants' swallowing function will be recorded, and the evaluators will be blinded to treatment at the assessment of the FEES.

Clinical data will be obtained from the participants' journal part 1 and 2 regarding sex, age, weight, height, body mass index (BMI), presence of a tracheostomy and if presence what type of tube used, length of intubation, presence of pneumonia, length stay at the hospital or ICU, medical diagnoses, the severity of the spinal cord injury according to the American Spinal Injury Association (ASIA) impairment scale, level of spinal cord injury and whether left or right approach was used during the ACSS will be recorded. Prior to the first assessment of the participant's swallowing function, written or oral (if tetraplegia) consent will be collected from each patient.

ELIGIBILITY:
Inclusion Criteria:

* All patients enrolled at the University Hospital of Umeå who have undergone ACSS between C2 and Th1 level due to trauma are eligible participants in the first part of the study.
* Eligibility criteria to participate in part 2 is swallowing dysfunction on FEES at 4±1-week post-operation

Exclusion Criteria:

* Patients <18 years of age
* known dysphagia prior to the trauma/injury
* affected brainstem that is shown on a CT or MRI
* severe brain damage.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-17 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Dysphagia severity | At start, at 4 weeks into the training, at end of treatment (after 8 weeks) and 12 ± 3 months post-intervention
  Change in swallowing function measured by FEES.

SECONDARY OUTCOMES:
Swallowing ability | At start, at 4 weeks into the training, at end of treatment (after 8 weeks) and 12 ± 3 months post-intervention
  Change in swallowing ability measured by the FOIS (functional oral intake scale)
Swallowing related quality of life | At start, at end of treatment (after 8 weeks) and 12 ± 3 months post-intervention
  Change in quality of life related to swallowing measured by the SWAL-QOL questionnaire.
Nutritional status | At start, at end of treatment (after 8 weeks) and 12 ± 3 months post-intervention
  Changes in nutritional status measured by the NRS-2002
Nutritional and metabolic status | At start, at end of treatment (after 8 weeks) and 12 ± 3 months post-intervention
  Changes in nutritional status measured by blood samples (i.e., levels of Albumin, levels of Leptin, Ghrelin and Adiponektin and also metabolites as ketone bodies)
The frequency of pneumonia | At start, at end of treatment (after 8 weeks) and 12 ± 3 months post-intervention
  The frequency of pneumonia will be will be registered and compared between the intervention and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Hägglund, PhD/SLP, Principal Investigator — Umeå University
Locations (1):
- University Hospital of Umeå, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No